CLINICAL TRIAL: NCT05706883
Title: Mutational Profile of Patients With and Without Neck and Supraclavicular Lymph Nodes Metastasis From Advanced Non-squamous Non-small-cell Lung Cancer: a Prospective Cohort Study
Brief Title: Clinical and Molecular Findings in Patients With Cervical/Supraclavicular Metastasis From Non-small-cell Lung Cancer (NSCLC)
Acronym: ProphetaPro
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5394
Record Dates: First submitted 2023-01-09; First posted 2023-01-31 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer Metastatic
MeSH Terms: interventions — Needles; Surgical Instruments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Patients with advanced lung cancer featuring cervical and/or supraclavicular lymph node metastasis
  Interventions: Procedure: Needle or forceps biopsy of cervical and/or supraclavicular lymph nodes
- Control group: Patients with advanced lung cancer NOT featuring cervical and/or supraclavicular lymph node metastasis
  Interventions: Procedure: Needle, forceps or surgical biopsy of any lesion other than cervical and/or supraclavicular lymph nodes

INTERVENTIONS:
Procedure: Needle or forceps biopsy of cervical and/or supraclavicular lymph nodes — Patients with evidence of enlarged and/or PET positive cervical and/or supraclavicular lymph nodes suspected of being metastasis from lung cancer will be submitted to the biopsy from this location.
  Other Names: Ultrasound guided biopsy
  Groups: Experimental group
Procedure: Needle, forceps or surgical biopsy of any lesion other than cervical and/or supraclavicular lymph nodes — Patients without evidence of enlarged and/or PET positive cervical and/or supraclavicular lymph nodes will be submitted to the biopsy considered less invasive and effective based on imaging data and clinical health status.
  Other Names: Ultrasound guided biopsy; Forceps biopsy during bronchoscopy; Surgical biopsy
  Groups: Control group

SUMMARY:
Despite the availability of highly effective endoscopy-based and computed tomography (CT)-based biopsy procedures, up to 50% of patients with advanced lung cancer potentially eligible for targeted therapies or immunotherapy do not have access to a diagnosis or to a thorough molecular profiling for different reasons. Enlarged and/or positron emission tomography (PET) positive cervical/supraclavicular lymph nodes (CSLs) are ideal targets for a minimally invasive diagnosis of lung cancer through a percutaneous ultrasound-guided biopsy (US-NAB). However, the prevalence of metastatic involvement of CSLs in patients with advanced lung cancer was never specifically assessed. Furthermore, the possible association of malignant CSLs involvement with molecular status was never investigated, unlike what was done for several other metastatic sites.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years at the time of the procedure;
* Suspected advanced, treatment naïve non-squamous NSCLC ;
* Indication to biopsy for diagnosis and/or molecular profiling;
* Written informed consent to the study participation.

Exclusion Criteria:

* Patients with known non-squamous NSCLC sent for re-biopsy after first or second line treatment;
* Inability to stop anticoagulant or antiplatelet therapy before the procedure (except acetylsalicylic acid 100 mg/day);
* Platelet count <50.000 per μL;
* Inability or unwillingness to provide a written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical and radiological suspicion of advanced lung cancer
Sampling Method: Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of KRAS mutation | 2 months
  Number of participants with KRAS mutation in the 2 groups (patients with and without cervical/supraclavicular lymph node metastasis)

SECONDARY OUTCOMES:
Prevalence of EGFR, ALK, ROS1, BRAF, RET, MET, NTRK | 2 months
  Number of participants with EGFR, ALK, ROS1, BRAF, RET, MET, NTRK mutation in the 2 groups (patients with and without cervical/supraclavicular lymph node metastasis)
Tumor proportion score of PD-L1 | 2 months
  Number of participants with a tumor proportion score of PD-L1 < 1%; 1-50%; >50% in the two groups (patients with and without cervical/supraclavicular lymph node metastasis)
Prevalence of cervical/supraclavicular lymph node metastasis | 2 months
  Number of participants with cervical/supraclavicular lymph node metastasis in the whole cohort of patients with stage IV lung cancer
Predictors of cervical/supraclavicular lymph node metastasis | 6 months
  Association between the presence of cervical/supraclavicular lymph node metastasis and the following factors: age, sex, smoking habit, tumor histologic type, central vs peripheral primary tumor, enlarged and/or PET positive N2 or N3 lymph nodes in the middle mediastinum, and molecular profile.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No